Ventilation **Noninvasive** for **Preterm Neonates** With Respiratory Distress Syndrome: a Multi-center Randomized **Controlled Trial** 

> (NCT03099694) 13 July 2017

Solid PDFIA EXPRESS COMP

#### STUDY PROTOCOL

Noninvasive high-frequency oscillatory ventilation versus nasal continuous positive airway pressure in preterm infants with respiratory distress syndrome: Study protocol for a multi-center, prospective, randomized, controlled trial. For the Noninvasive High-Frequency Oscillatory Ventilation Study Group (NHFOV Study Group\*).

#### **Abstract**

Background: Invasive mechanical ventilation it associated with development of adverse pulmonary and non-pulmonary outcomes in very low birt's weight infants. Various modes of non-invasive respitatory support are being increasingly used to decrease the incidence of brought pulmonary dysplasia (EPD). The aim of this trial is to compare the effect of noninvasive high-frequency oscillatory ventilation (NHFOV) and nasal continuous positive airway pressure (NCPAP) in preterm infants with respiratory distress syndrome (RDS) as a primary noninvasive ventilation support mode.

Methods/Design: In this multicenter, randomized, controlled trial, 300 preterm infants born at gertational age (GA) less than 34 weeks with a diagnosis of RDS will be randomized to NHFOV or NCPAP as a primary mode of noninvasive respiratory suprem. Study will be conducted in 18 tertiary neonatal intensive care units in China. The primary outcome is the need for invasive mechanical ventilation (IMV) during the first 7 days after enrollment in preterm infants randomized to the two groups. The



prespecified secondary outcomes include days of hospitalization, days on noninvasive respiratory support, days on IMV, days on supplemental oxygen, mortality, need for surfactant, severe retinopathy of prematurity(ROP) requiring laser or surgery, patent ductus arteriosus needing ligation, bronchopulmonary dysplasia(BPD), occurrence of abdominal distention, air leaksyndromes, intraventricular hemorrhage (IVH ≥ grade 3), necrotizing enterocolitis (NEC> II stage) and nasal trauma. Other secondary outcomes include Bayley Scales of Infant Development at 18-24 months of corrected age.

Trial registration: ClinicalTrials.gov Identifier: NC 03099694.

Key words: Noninvasive high-frequency oscillatory ventilation; nasal continuous s syndro

s syndro

the syndro

the syndro positive airway pressure; respiratory distress syndrome; proterm infants; surfactant; invasive mechanical ventila, on



## **Background**

Respiratory distress syndrome (RDS) due to surfactant deficiency is the leading cause of respiratory failure in preterm infants [1]. Early noninvasive positive pressure ventilation has become a recommended strategy for respiratory management of preterm infants with RDS [2]. In addition to nasal continuous positive airway pressure (NCPAP), various types of noninvasive ventilation(NIV) modes have been used in the treatment of RDS including heated, humidified, high-flow nasal cannula (HHFNC), biphasic NCPAP (BP-NCPAP) and nasal intermittent positive airway pressure(NIPPV) [3]. However, clinical trials have shown that 25 to 6700sf very low birth weight preterm infants fail these NIV modes and require 1.1V [4-5]. To minimize the need of IMV, noninvasive high-frequency oscilla ry ventilation (NHFOV) has been studied as a rescue treatment after failure of o her NIV modes or fol owing extubation from IMV during weaning phase [6]. However, to date, no studies have been published on the efficacy of NHFOV as a primary mode of raphatory support in preterm infants. In the present that we aim to compare the effect of NHFOV and NCPAP in preterm infants with RDS as a primary NIV mode. Our main hypothesis is that NHFOV is more effective in the treatment of preterm infants with RDS than NCPAP when used as a primary NIV mode

## **Trial Design**

#### Aim

The primary aim of this trial is to compare the need for IMV during the first 7 days of life in infants randomized to NHFOV versus NCPAP.

#### Study design

This will be a multi-center, prospective, randomized controlled trial conducted in 18 tertiary neonatal intensive care units (NICUs) in China. The trial will be performed in accordance with prospective trial flow (Fig.1).

#### **Inclusion criteria:**

(1) Gestational age (GA) is from 26 weeks 0 days (26<sup>+0</sup>weeks) to 33 weeks 6 days(33<sup>+0</sup>weeks) (estimated on the postmenstrual date and early gestation ultrasonographic findings); (2) diagnosis of RDS. The diagnosis of RDS will be based on clinical manifestations(tachypnea, nasal flaring and or grunting) and the typical X-ray picture of RDS (grain shadow, air bronchography white lung)-see appendix; (3) RDS Silverman score>5; (4) Age <12 hours: (5) informed parental consent has been obtained.

#### **Exclusion criteria**

(1) Resuscitation requiring early intubation according to the American Academy of Pediatrics guidelines for neonatal resuscitation [8]; (2)major congenital malformations of known complex congenital heart disease; (3)pulmonary hemorrhage or pneumothorax; (4) congenital lang diseases or malformations or pulmonary hypoplasia;

#### **Setting**

We plan to entail preterm infants born between 26 and 34 weeks of gestational age from 15 te. dary NICUs in China. These 18 tertiary NICUs have more than 800 NICU beds and annual admissions of nearly 8,000 preterm infants with RDS each year. The first (XZ) and last authors (RR) take responsibility for the accuracy and completeness



of the trial.

#### Randomization

To avoid the chance of having more infants in one group than another, block randomization will be applied, with a block size of 4. The envelopes are sealed, shuffled, and then numbered in sequential order from 1 to 4. A clinician who is not in the trial group will open the envelope and randomize patients. This procedure will be repeated for each group of four infants. Infants will be stratified according to  $26^{0/7}$ - $27^{6/7}$ weeks,  $28^{0/7}$ - $29^{6/7}$ weeks,  $30^{0/7}$ - $31^{6/7}$  weeks and  $32^{0/7}$ - $33^{6/7}$ weeks. Infants born from multiple gestations will be assigned by in Jividual randomization. Infants randomized to one arm cannot crossover to the other or vice-versa during the study.

#### **Trial intervention**

#### Ventilators

CPAP: CPAP will be provided by continuous row devices (CNO Medin, Germany or Carefusion, USA) Bubble CPAP devices will not be used.

NHFOV: NHTOV will be provided by two ventilators (CNO, Medin, Germany or SLE 5000, UK). The Medin CNC ventilator produces high-frequency oscillations by flow interruption with cyclic opening-closure of the end expiratory valve. Otherwise, The SLE 5000 ventilator is a fine-cycled, pressure-limited and continuous-flow neonatal ventilator.

Before the teaming of the study all ventilators will be checked to ensure that there is no malfunction

#### Interfaces

CPAP and NHFOV will be all administered through short, low-resistance binasal prongs,



since these are supposed to be the best in terms of resistive charge, leaks and/of comfort. Nasal prongs size will be chosen according to the nares' diameter as the best fitting ones (the largest ones that fit the nares without blanching the surrounding tissues) and following manufacturer's recommendations. Particular care (e.g.: pacifiers, positioning, nursing) will be applied to reduce leaks and improve patients' comfort. These latters will be evaluated through a dedicated 30 min observation period when study intervention will be instigated.

### Ventilatory management

The two different respiratory supports will be managed as follows:

CPAP: Neonates assigned to the CPAP group vere initiated on a pressure of 5 cmH<sub>2</sub>O. CPAP can be raised in steps of 1 cmH<sub>2</sub>O to 10 cmH<sub>2</sub>O. If this is not enough to maintain target oxygen saturatio (SpO<sub>2</sub>) from 89% to 92% in preterm infants <30 weeks GA and 90-94% in intants ≥30 weeks GA by ruise oximeter, FiO<sub>2</sub> will be added up to 0.40.

PNHFOV: For Media CNO, the initial NHFO settings will be: mean airway pressure (MAP) of 6cmH<sub>2</sub>O(range 5-10cmH<sub>2</sub>O), frequency of 10 Hz(range 6-12), The Media CNO has fell grades of amplitude, grade 7th amplitude will be to start with (grade range 7th-10th). For SLE 5000, The initial settings will be: MAP of community community frequency of 10Hz (range 6-12), inspiratory time 50% (1:1), oscillations of amplitude of 20 cm H<sub>2</sub>O(range 6-12), inspiratory time 50% (1:1), oscillations of amplitude of 20 cm H<sub>2</sub>O(range 6-12). It is not strictly necessary to have visible chest oscillations, as most of the CO2 elimination during NHFOV will occur in the upper airway dead space. Maximal allowed FiO<sub>2</sub> will be 0.40 and SpO<sub>2</sub> from 89% to 93% in



preterm infants <30 weeks GA and 90-94% in infants ≥30 weeks GA by pulse oximeter.

### **Surfactant Therapy**

Surfactant (Poractant alfa, Chiesi Pharmaceuticals, Parma, Italy) at dose of 200 mg/kg will be administered via INSURE method if infant presents with the following: infants≤26 week's gestation when FiO<sub>2</sub> requirement >0.30 and infants>26 week's gestation when FiO<sub>2</sub> requirement >0.40 [2]. Additional doses of surfactant may be given using INSURE technique at the discretion of the clinician.

### **Caffeine Therapy**

Caffeine (Caffeine Citrate Injection. Chiesi I ha maceuticals, Parma, Italy) will be administered when infants present with moderate apnea (defined as 3 or more episodes in 24 hours or a single episode requiring respectation and bag-mask ventilation). The initial loading dose is 20mg/kg, an take maintenance dose is 5mg/kg per day.

# Weaning from study interventions

The criteria for weaning nonin (a.1) respiratory will be: (1) minimal or no signs of respiratory distress (RDS Si verman score < 5); (2) NHFOV MAP or NCPAP pressure <6cmH<sub>2</sub>O 21.1 (3) FiO<sub>2</sub><0.25 to achieve target SpO<sub>2</sub>.

### Criteria for intubation and IMV

These win be as follows [10-11]: (1) severe respiratory acidosis ( $P_aCO_2>65$  mmHg with pH<7.20);(2) severe apnea and bradycardia (defined as recurrent apnea with >3 episodes per hour associated with heart rate < 100/min, a single episode of apnea that



requires bag and mask ventilation); (3)hypoxia (FiO<sub>2</sub>>0.5 with PaO<sub>2</sub><50mmHg), severe respiratory distress (RDS Silverman score > 7); (4) pulmonary hemorrhage; (5) pneumothorax; (6) cardiopulmonary arrest needing chest compressions.

### Training

Since not all clinicians are well versed in all respiratory techniques and, particularly, NHFOV is a relatively new technique, the training is capital for the trial success. The protocol will be diffused between participating centers at least 3 months before the study begins. One investigator (YS) will explain the study protocol in an in-person meeting with all investigators. During the two months' period, clinicians will familiarize with the protocol and  $\hat{u}$  respiratory techniques and the two co-principal investigators will be available to solve up doubt. A dedicated social media chat has been set to facilitate these exchanges. The trial is supposed to actually furthin July 2017.

#### **Outcomes**

The primary outcome of this trial will be to determine the first 7 days of life in preterm infants randomzed to the two groups. Secondary outcomes include days of hospitalization, days on noninvasive vertication, days on supplemental oxygen, predischarge mortality, surfactant doses, incidence and stage III ROP and BPD, occurrences of abdominal distention, air leaks, IVH  $\geq$  grade 3 and NEC. Secondary outcomes also include Bayley Scales of Infant Development at 18-24 months of corrected age. BPD will be defined according to the National Institutes of Health consensus definition as mild, moderate and severe BPD [12], IVH classification according to Papile et al [13] and for NEC, Bell staging will be used [14].

#### **Data collection**

Patient demographic data include: sex, birth weight, gestational age, Apgar scores, mode of

delivery, prenatal corticosteroid use, premature rupture of the membrane, RDS Silverman score and critical risk index for babies-II (CRIB-II) score. More details see in the appendixClinical data:Including the need for IMV, days of hospitalization, days on noninvasive respiratory support, days on supplemental oxygen, mortality, the need for surfactant, occurrences of abdominal distention, air leaks, IVH ≥ grade and NEC≥stage II. More details see in the appendixFollow-up data: The incidence of BPD and ROP at a post-menstrual age of 36 weeks or at discharge, and Bayley Scales of Infant Development at 18-24 months of corrected age.

### Sample size calculation

It is difficult to calculate a sample size for such a study, since it is the first to investigate NHFOV vs CPAP in primary support phase in preterm infacts with RDS. There is only one preliminary study available about the primary outcome "need for IMV". This pilot study conducted by Zhu et al provides data about the primary outcome "need for IMV". This trial showed the need for IMV was significantly lower in the NHFOV compared with the NCPAP group (24.3% vs. 56.4%, P<0.01). Considering an arriverror of 0.05 and a power of 90%, 150 neonates should be enrolled in each arm (with a 1:1 design) to detect the same difference.

### Statistical methods

Data will be analyzed using SPSS version 19 software. The statistical analyses include Student's test for continuous data and compared proportions using Chi-squared test, and Fisher's exact test for categorical data. Predefined four subgroups are  $26^{0/7}$ - $27^{6/7}$ weeks,  $28^{0/7}$ - $29^{6/7}$ weeks,  $30^{0/7}$ - $31^{6/7}$  weeks and  $32^{0/7}$ - $33^{6/7}$ weeks, and subgroup analyses will be conducted for the primary outcome in the preterm infants. To further evaluate the effect of NHFOV on intubation within



subgroup, the test of treatment-by-gestational age subgroup interaction will also be done using the paired binary logistic regression. For the preterm infants lost to follow-up, the missing values of the primary and secondary outcomes are replaced using multiple imputation. A P-value < 0.05 will be regarded as statistically significant.

Data Safety Monitoring Board (DSMB): Dr. Kris Sekar, Professor of Pediatrics, Oklahoma University Medical Center, Oklahoma, Dr. Jatinder Bhatia, Professor of Pediatrics, Medical College of Georgia, Georgia Health Sciences University, Augusta, Georgia, and Dr. Rowena Cayabyab, MD., MPH Destatistics and Epidemiology) Assistant Professor of Pediatrics, Keck School of Medicine of the University of Southern California, Los Angeles, California will serve as PSMB members. Dr. Cayabyab will also serve as control and for statistical analysis.

### Registration number

The trial has been approved by the centralized ethics committee (The Ethics Committee of Daping Hospital, Research institute of Surgery, Third Military Medical University) and registered at <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>(ID: NCT03099694).

#### **Discussion**

In the past decades, several clinical trials have compared the effects between NHFOV and NCPAP in reconates as a rescue mode or during weaning from IMV. These trials demonstrated that NHFOV applied with nasopharyngeal tube are more beneficial than NCPAP in reducing CO<sub>2</sub> levels [16-19]. Recently, two retrospective case series also reported NHFOV could be applied in preterm infants as a rescue treatment after the



failure of other noninvasive ventilation modes[15,20]. However, there are some limitations in these trials: 1) small sample size; 2) lack of a prospective, randomized trial design; and 3) wide range of NHFOV parameters used in these trials. Given these limitations, a multi-center, prospective, randomized, controlled trial is necessary for better evaluation of NHFOV as a primary mode of noninvasive support. To our knowledge, this will be the first multi-center prospective randomized controlled trial for evaluation of NHFOV as a primary noninvasive mode in preterm infants with RDS in China or any other part of the world. Our trial may help contribute to establish guidelines for NHFOV in preterm infants with RD5 to minimize the need for IMV, and to decrease significant pulmonary and non pulmonary morbidities associated with IMV.

#### **Funding**

The trial is initiated and planned by the researchers and funded by Scientific Research Projects unit of Changing (Project-cstc2016sh.ns-ztzx13001)

### Acknowledgement

The authors would like to thank all families whose infants will participate in this trial, and staff providing patient care in all the participating sites.

### **Conflict of Interest**

None of the where have declared conflicts of interests to participate in this trial.

#### **APPENDIX**

#### A1. Diagnosis of RDS:

Respiratory distress appearing within the first 24 h of life, with complete, sustained, and prompt response to surfactant or lung recruitment orboth; additional non-mandatory criteria are



lung imaging (chest X-rays or ultrasound, according to local policies) supporting the diagnosis or lamellar body counts \le 30 000/mm³, or both

#### A2. CLARIFICATIONS FOR EXCLUSION CRITERIA

Some exclusion criteria are represented by congenital disorders: when a patient is affected by these disorders his biology and physiology are significantly changed and are not eligible for the study and will not be randomized. If the condition has been discovered/suspected after the randomization but before the study inclusion (that is, before extubation), they will not receive the study intervention and will not entry in the study. If one of these conditions is diagnosed after the inclusion in the study, the neonate will be excluded *a posteriori*. This is the case of neonates withmajor congenital anomalies, chromosomal abnormalities auromuscular diseases, congenital upper respiratory tract abnormalities and congenital lung. Jiseases or malformations or hypoplasia. Examples of these conditions are: genetic syndromes, surfactant protein defects, congenital adenomatous pulmonary malformations, congenital diaphragmatic hermin or sequestration, congenital hypoventilation syndromes, pulmonary hypoplasia or any metabolic disease.

# A3. LIST OF STUDY DEFINIT: ON

- or early ultrasound scan (within the first trimester). If a discrepancy of more than 2 weeks exists, the early ultrasound scan will be chosen.
- **INSURE.** Intubation—Syrfactant-Extubation
- Antenatal stere is: Antenatal steroid prophylaxis will be considered complete if two 12 mg assess of betamethasone 24h apart and between 1 day and 7 days before the delivery had been given.
- Clinical Risk Index for Babies (CRIB-II) score. This is an estimator of the clinical severity at the NICU admission. CRIB-II score considers 4 variables: birth weight, GA, base excess within the 1sthour of life and temperature at



theadmission(see below). An online calculator is available at www.sfar.org/scores2/crib22.php



- Premature rupture of the membrane. Premature unture of the membrane will be considered complete it more than 18 hours.
- **Abdominal distriction.** Abdominal circumference (cm) at 48h and 96h after study intervention.

#### References

- 1. Mathal SS, Raju U, Kam Lkar M. Management of respiratory distress in the newborn. Med J Armed Forces India 2007; 63: 269-272.
- 2. Sweet DG. Ca nielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, et al. European consensus guidelines on harnanagement of respiratory distress syndrome-2016 update.

  Neonatology2017;111:107-125.
- 3. Cumming JJ, Polin RA, AAP the COMMITTEE ON FETUS AND NEWBORN. Noninvasive respiratory support. Pediatrics2016; 137(1):

- e20153758. http://dx.doi.org/doi: 10.1542/peds.2015-3758.
- 4. Stefanescu BM, Murphy WP, Hansell BJ, Fuloria M, Morgan TM, Aschner JL. A randomized, controlled trial comparing two different continuous positive airway pressure systems for the successful extubation of extremely low birth weight infants. Pediatrics2003; 112:1031–1038.
- Barrington KJ, Bull D, Finer NN. Randomized trial of nasal synchronized intermittent mandatory ventilation compared with continuous positive airway pressure after extubation of very low birth weight infants. Pediatrics2001; 107:638–641.
- 6. Ramanathan R, Sekar KC, Rasmussen M, Bhatia J, Soll RF. Nasal intermittent positive pressure ventilation after surfactory treatment for respiratory distress syndrome in preterm infants <30 v ecks gestation: a randomize it, controlled trial. J Perinatal 2012;32:336 3:15
- 7. Fischer HS, Bohlin K, Bull of C, Schmalisch G, Chemer M, Reiss L, Czernik C. Nasal high-frequency oscillation ventilation in neonates: a survey in five Europeancountries. Eur J Pediatr2015:174, 465-471.
- 8. Perlman M, Wyllie J, Kattwinke J. Atkins DL, Chameides L, Goldsmith JP, Guinsburg R, Hazinski MF Morley C, Richmond S, et al. Neonatal Resuscitation Chapter Collaborators. Part 11: Neonatal resuscitation: 2010 International Contensus on Cardiopulmonary Resuscitation And Emergency Cardiovascular Care Science With Treatment Recommendations.

  Circumtion2010; 122(16)(suppl2):S516-S538.
- 9. Czyabyab R, Arora V, Wertheimer F, Durand M, Ramanathan R. Graded oxygen saturation targets and retinopathy of prematurity in extremely preterm infants. Pediatric Research 2016;80:401-406.



- 10. Lista G, Casoldi F, Fotana P, Daniele L, Caviqioli F, Rossi S, Mancuso D, Reali R. Nasal continuous positive airway pressure (CPAP) versus bi-level nasal CPAP in preterm babies with respiratory distress syndrome: a randomized control trial. Arch Dis Child Fetal Neonatal Ed, 2010;95:F85-F89.
- 11. O'Brien K, Campell C, Brown L, Wenger L, Shah L. Infant flow biphasic nasal continuous positive airway pressure (BP-NCPAP) vs. infant flow NCPAP for the facilitation of extubation in infants≤1,250 grams: a randomized controlled trial. BMC Pediatr2012; 12: 43-51.
- 12. Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J RespirCrit Care Med 2001; 163: 1723-1729.
- 13. Papile LA, Burstein J, Burstein R, Koffler M. Incidence and evolution of subependymal and intraventricular temorrhage: a study of in ants with birth weights less than 1,500gm J Pe tiatr1978; 92: 529-534
- 14. Bell MJ, Ternberg JL, Feis in RD, et al. Neonatal necrotizing ebterocolitis: therapeutic decisions based upon clinical stocing. Ann Surg 1978;187:1-7.
- 15. Wang CH, Sh. LP, Ma XL, Lin HJ, Xv YP, Du LZ. Use of noninvasive high-frequency oscillatory vertibation in very low birth weight infants.

  ZhonghuaErKeZaZhi 2017, 5): 177-181.
- 16. Van der Hoeven M. Prouwer E, Blanco CE. Nasal high frequency ventilation in neonates with a oderate respiratory insufficiency. Arch Dis Child Fetal Neonatal 1.1 1998; 79(1): F61–F63.
- 17. Colaizy TT, Younis UM, Bell EF, Klein JM. Nasal high-frequency ventilation for premature infants. Acta Paediatr 2008; 97: 1518–1522.
- 18. Czernik C, Schmalisch G, Bührer C, Proquitté H. Weaning of neonates from mechanical ventilation by use of nasopharyngeal high frequency oscillatory



- ventilation: a preliminary study. J Matern Fetal Neonatal Med2012; 25: 374-378.
- 19. Aktas S, Unal S, Aksu M, Ozcan E, Ergenekon E, Turkyilmaz C, Hirfanoglu L, Atalay Y. Nasal HFOV with Binasal Cannula appears effective and feasible in ELBW Newborns. J Trop Pediatr 2016; 62: 165-168.
- 20. Mukerji A, Singh B, Helou SE, Fusch C, Dunn M, Belik J, Shah V. Use of noninvasive high frequency ventilation in the neonatal intensive care unit: a retrospective review. Am J Perinatol2015; 30: 171-176.http://dx.doi.org/doi:

